CLINICAL TRIAL: NCT01352312
Title: Phase I Trial With Cohort Expansion of Pentostatin, Bendamustine and Ofatumumab (PBO) for the Treatment of Chronic Lymphocytic Leukemia and Non-Hodgkin's Lymphoma
Brief Title: Combination of Pentostatin, Bendamustine and Ofatumumab for Treatment of Chronic Lymphocytic Leukemia and Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual over 12 mo period
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11P.166; 2011-23 (Other: CCRRC); OFT114197 (Other: GlaxoSmithKline); JT 1680 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; B-Cell Non-Hodgkin's Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma; B-cell; leukemia; lymphoma; bendamustine; pentostatin; ofatumumab; NHL; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma | interventions — Bendamustine Hydrochloride; Pentostatin; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pentostatin, bendamustine, ofatumumab) (Experimental): Patients receive bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, pentostatin IV on day 1, and ofatumumab IV on day 2. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine; Drug: Pentostatin; Drug: Ofatumumab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine at the dose of 50 mg/m2 (or 70 or 90 or 40 mg/m2 depending on the dose level) daily on day 1 and 2.
  Other Names: Ribomustin; Treanda; SDX-105
Drug: Pentostatin — Pentostatin 4 mg/m2 on day 1 of each cycle. For patients with estimated or measured glomerular filtration rate (GFR) 30 to 60 ml/min/m2 pentostatin will be administered at the reduced dose of 2 mg/m2 on day 1 of each cycle.
  Other Names: deoxycoformycin
Drug: Ofatumumab — Ofatumumab 300 mg on day 2 of first cycle. Subsequently, from cycle 2 to 6, ofatumumab 1000 mg on day 2 will be administered.
  Other Names: Arzerra; HuMax-CD20

SUMMARY:
This is a Phase 1 study with Cohort Expansion of Pentostatin, Bendamustine and Ofatumumab (PBO) for patients with previously treated Chronic Lymphocytic Leukemia (CLL) and B-cell Non-Hodgkin's Lymphoma (B- cell NHL). The purpose of this study is to determine the optimal dose of bendamustine in combination with pentostatin and ofatumumab, and then to see how safe these three drugs work together.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common form of leukemia in the United States. There has been considerable progress in understanding the biology and treatment of CLL in the last 20 years. However, even with modern therapies, complete responses (CR) are achieved in approximately 25% of the patients with relapsed/refractory disease. Multiple studies have demonstrated that patients who achieve CR have better clinical outcomes than patients who do not achieve a CR with therapy. B-cell NHL is composed of multiple subtypes of neoplasm. These diseases are closely related to CLL in terms of natural history, biology, and responsiveness to similar therapeutic agents. These diseases are not usually cured by available chemotherapy and ultimately patients succumb to progression of resistant disease. Therefore, there is a need to develop better therapies to improve survival in patients with CLL and B-cell NHL.

Preclinical and clinical data suggests that pentostatin, bendamustine, ofatumumab are active drugs for the treatment of B-cell malignancies. In an earlier clinical trial conducted by Dr. Weiss (lead site PI), the combination of pentostatin and cyclophosphamide had very good activity in previously treated patients with B-cell neoplasms. This regimen was also better tolerated than similar fludarabine-based regimen. The response rates were improved with addition of rituximab, anti CD 20 antibody, to the above regimen. Studies have demonstrated synergy between bendamustine and purine analogs like pentostatin in killing cancer cell types of CLL and NHL. The combination of these three drugs (pentostatin, bendamustine and ofatumumab) has not been tested in clinical setting and we anticipate that the combination regimen will be more active than individual drugs alone. The aim of this trial is to find a safe dose of bendamustine to be used in combination with pentostatin and ofatumumab in patients with previously treated CLL and B-cell NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated CLL or other B-cell neoplasm including small lymphocytic lymphoma, hairy cell leukemia, follicular, lymphoma, Waldenstrom's macroglobulinemia, marginal zone lymphomas, mantle cell lymphomas, lymphoplasmacytic lymphoma and diffuse large B-cell lymphoma. Patients with composite lymphoma and transformed disease will be included. Immunophenotypic (or immunohistochemical) analysis of the malignant lymphocytes should demonstrate that the cells are B-cells.
2. Patients must have had prior cytotoxic therapy for their disease. Patients with diffuse large B-cell lymphoma must have been treated with at least 2 prior cytotoxic therapies.
3. Age ≥ 18 years of age.
4. ECOG performance statue 0 to 2.
5. Reasonable life-expectancy greater than 12 weeks.
6. Patients with autoimmune hemolytic anemia or autoimmune thrombocytopenia will be eligible for treatment.
7. Signed informed consent, which indicates the investigational nature of this study, is required.
8. No patient may be entered onto the study without consultation with the principal investigator or his designee.

Exclusion Criteria:

1. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
2. No prior cytotoxic therapy for at least 4 weeks before enrollment.
3. Currently participating in any other interventional clinical study.
4. Other currently active malignancy.
5. Active uncontrolled infection.
6. History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
7. Known HIV positive.
8. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and uncontrolled symptomatic arrhythmia.
9. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
10. Positive serology for hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
11. Active hepatitis C infection. If positive serology for hepatitis C (HC) defined as a positive test for HCAb, HC quantitative PCR will be performed. If PCR is positive the subject will be excluded
12. Screening laboratory values:

    1. creatinine > 2.0 times upper normal limit and creatinine clearance < 30 ml/min/m2. Patients with creatinine > 2 times upper limit of normal will have creatinine clearance estimated. At the discretion of treating physician, creatinine clearance can be measured and that value can be used instead of calculated creatinine clearance.
    2. total bilirubin > 2 times upper normal limit (unless due to tumor involvement of liver or a known history of Gilbert's disease)
    3. ALT (alanine transaminase) > 2.5 times upper normal limit (unless due to disease involvement of liver.
13. Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
14. Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
15. Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Bendamustine | Up to 6 months
  The primary objective of this study is to determine the dose of bendamustine in combination with pentostatin and ofatumumab at which <33% of patients with relapsed Non-Hodgkin's Lymphoma (NHL) or Chronic Lymphocytic Leukemia (CLL) experience severe toxicity; and to assess the toxicity of this regimen.
Dose Limiting Toxicity (DLT) | Through one year post-treatment
  Dose limiting toxicity (DLT) will be defined as any grade 4 infection, or grade ≥ 3 non-hematologic toxicity that persists for 7 days or more.
  Safety Issue?: (FDAAA) Yes

SECONDARY OUTCOMES:
Efficacy of Study Treatment Regimen | 3 and 6 months
  1. CBC (complete blood count)
  2. B-cell count
  3. If a patient is in CR (complete recovery) by other criteria then bone marrow aspiration/biopsy will be performed.
  4. CT (x-ray computed tomography) scan of chest/abdomen/pelvis (optional in patients with CLL)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Fili, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org